CLINICAL TRIAL: NCT06821932
Title: Evaluation of the Bone Structure Surrounding Photofunctionalized Implants Using the Fractal Analysis Method: A Split-mouth Randomised Clinical Trial
Brief Title: Evaluation of the Bone Structure Surrounding Photofunctionalized Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Fatma Karacaoğlu, Assoc. Prof., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36290600/34/2021
Record Dates: First submitted 2025-01-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2021-04

CONDITIONS: Dental Implants
Keywords: Photofunctionalization; Ultraviyolet Light; Dental implant

STUDY DESIGN:
Intervention Model Description: Splith mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: photofunctionalized implant inserted (Experimental): Dental implants were subjected to the photofunctionalization process and then immediately inserted into the bone on the experimental side of the mouth
  Interventions: Procedure: Photofunctionalized dental implant surgery
- Control: Dental implant placement without photofunctionalization process (Active Comparator): Dental implants were inserted in the bone on the contralateral side of the mouth without photofunctionalization
  Interventions: Procedure: Dental implant surgery

INTERVENTIONS:
Procedure: Photofunctionalized dental implant surgery — Dental implants subjected to photofunctionalization were placed in the experimental area of the mouth.
  Arms: Experimental: photofunctionalized implant inserted
Procedure: Dental implant surgery — Dental implants not subjected to photofunctionalization were placed in the bone on the contralateral side of the mouth
  Arms: Control: Dental implant placement without photofunctionalization process

SUMMARY:
Bacground: Implant failure may necessitate the need for another surgical procedure to improve implant survival. Photofunctionalization with UV is a practice that can positively affect dental implant success and osseointegration. The aim of this study is to evaluate the effect of the photofunctionalization process on the bone quality around the implant.

Methods: In the study, 42 implants were evaluated using the Fractal Analysis method from the panoramic radiographs taken before and after the implant. The analysis of the data was done with the SPSS 26 program and worked with a 95% confidence level. In the test group, there was a statistically significant difference between the 1st panoramic measurement and the 2nd panoramic measurement (p=0.044<0.05) and the bone fractal score increased.

DETAILED DESCRIPTION:
Bacground: Implant failure may necessitate the need for another surgical procedure to improve implant survival. Photofunctionalization with UV is a practice that can positively affect dental implant success and osseointegration. The aim of this study is to evaluate the effect of the photofunctionalization process on the bone quality around the implant.

Methods: In the study, 42 implants were evaluated using the Fractal Analysis method from the panoramic radiographs taken before and after the implant. The analysis of the data was done with the SPSS 26 program and worked with a 95% confidence level. In the test group, there was a statistically significant difference between the 1st panoramic measurement and the 2nd panoramic measurement (p=0.044<0.05) and the bone fractal score increased.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Having bilateral edentulous areas in the posterior mandibular region

Exclusion Criteria:

* Individuals with any systemic disease,
* Individuals using drugs that affect bone metabolism,
* Patients with findings that could affect the study results such as bone cysts, tumors, lesions or fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Bone fractal analysis | 1 month
  The bone fractal dimension (FB) values were determined by sizing the ROI to 25x25 pixels using the box counting method. The area of interest to be examined in the image was cropped and saved in 8-bit format. Different image processing methods were applied. For the fractal dimension calculation the box counting method was used. The number of squares containing trabeculae and the total number of squares in the image were determined for various pixel sizes. These values were plotted on a logarithmic scale, and the slope of the line that best fit the points on the graph determined the bone FB.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choi B, Lee YC, Oh KC, Lee JH. Effects of photofunctionalization on early osseointegration of titanium dental implants in the maxillary posterior region: a randomized double-blinded clinical trial. Int J Implant Dent. 2021 May 10;7(1):37. doi: 10.1186/s40729-021-00318-x. PMID 33969450
- [Background] Hirota M, Ozawa T, Iwai T, Ogawa T, Tohnai I. Effect of Photofunctionalization on Early Implant Failure. Int J Oral Maxillofac Implants. 2018 Sep/Oct;33(5):1098-1102. doi: 10.11607/jomi.6541. PMID 30231097
- [Derived] Farsiani H, Bagis N, Balkan EP, Karacaoglu F, Guner ZD, Orhan K. Evaluation of the bone structure surrounding photofunctionalized implants using the fractal analysis method: a split-mouth randomized clinical study. BMC Oral Health. 2025 Jul 1;25(1):964. doi: 10.1186/s12903-025-06330-6. PMID 40598042